CLINICAL TRIAL: NCT03365258
Title: The Effect of Applying Modified NUTRIC Scoring System to Evaluate the Nutrition Risk and Giving Different Types of Nutritional Support on Clinical Outcomes in Critically Ill Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, Wang, Chen-Yu, Director of Medical Intensive Care Unit, Taichung Veterans General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CF17249A
Record Dates: First submitted 2017-11-28; First posted 2017-12-07 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Nutritional Risk (Other): modified NUTRIC score ≥ 5
  Interventions: Dietary Supplement: Trophic feeding; Dietary Supplement: volume-based feeding
- Low Nutritional Risk (Other): modified NUTRIC score < 5
  Interventions: Dietary Supplement: Trophic feeding; Dietary Supplement: volume-based feeding

INTERVENTIONS:
Dietary Supplement: Trophic feeding — Non-blind to randomize to trophic feeding group and volume based feeding group in the first six days (Day 0->Day 6). The definition of trophic feeding is continue feeding with feeding rate: 20 kcal/hr.
Dietary Supplement: volume-based feeding — Non-blind to randomize to trophic feeding group and volume based feeding group in the first six days (Day 0->Day 6). The definition Volume-based feeding also use continue feeding by feeding protocol
  Other Names: Full caloric feeding

SUMMARY:
Malnutrition is very common in critically ill patients. It is quite important to evaluate nutritional status precisely. Heyland et al firstly reported NUTRIC score including age, APACHE II score, SOFA score, number of commorbidities, days from hospital to ICU admission and IL-6. Because the IL-6 is not routinely checked at ICU. A modified NUTRIC score without IL-6 is more practical. Previous studies showed lower in-hospital mortality in higher nutritional risk patients with higher caloric intake compared with lower caloric intake. However, there is still controversial regarding the in-hospital mortality between full caloric feeding and permissive underfeeding in critically ill patients. Herein the investigators conduct a study to investigate what kinds of nutritional supplements will decrease in-hospital mortality in different nutritional risk patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Medical intensive care unit patients 2. age elder than 20 years old 3. Intubated with ventilator support patients 4. Predicted ICU stay longer than 72 hours

Exclusion Criteria:

* 1. NPO patients 2. Contraindication for enteral feeding 3. TPN use 4. Upper or lower GI bleeding patients 5. Feeding with gastrostomy or Jejunostomy patients 6. Metoclopramide related EPS or Torsades de pointes history

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-12-28 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | 90 days
  mortality or discharge

CONTACTS AND LOCATIONS:
Locations (1):
- 王振宇, Taichung, 台中市, Taiwan